CLINICAL TRIAL: NCT04685395
Title: Comparative Efﬁcacy of Rebamipide Gargle And Benzydamine HCL Gargle in Prevention and Management of Chemo- and Radio-therapy-induced Oral Mucositis in Head and Neck Cancer Patients: (A Randomized Clinical Trial)
Brief Title: Comparative Efﬁcacy of Rebamipide Gargle And Benzydamine HCL Gargle in Prevention and Management of Chemo- and Radio-therapy-induced Oral Mucositis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Belag, assisstant lecture, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OMED2-2-1
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: Parallel group, two arm, superiority randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benzydamine hydrochloride (Active Comparator): group I ( benzdymine HCL ); subject will be instructed to use Benzydamine hydrochloride gargle 6 times daily and not to eat or drink for the subsequent 10 min from first day of radiation therapy (4-6 week) until 2 weeks after the end of treatment(end of radiation ).
  dose :5 ml every time dosage form ; mouth wash
  Interventions: Drug: Ribamipide gargle \benzdymine HCL gargel
- Rebamipide (Active Comparator): group II ( rebamipide) :subject will be instructed to use Rebamipide gargle 6 times daily and not to eat or drink for the subsequent 10 min from first day of radiation therapy (4-6 week) until 2 weeks after the end of treatment(end of radiation ).
  dosage form ; mouth wash
  Interventions: Drug: Ribamipide gargle \benzdymine HCL gargel

INTERVENTIONS:
Drug: Ribamipide gargle \benzdymine HCL gargel — ribamipide gargle 6 time daily 5ml dosage
  Other Names: Ribamipide gargle \tantum mouth wash

SUMMARY:
evaluate preventive and therapeutic effects of Rebamipide gargle on reducing incidence of oral mucositis in comparison with benzydamine HCL mouthwash.

DETAILED DESCRIPTION:
Oral mucositis is a common and potentially dangerous complication of anticancer treatment. Inflammation and ulcerations of the oral mucosa make swallowing and, thereby, eating and drinking, difficult or even impossible, leading to anorexia and weight loss(Araújo et al., 2018) .There is a serious risk of infections and even sepsis, particularly in immune-ompromised patients. OM is associated with severe pain, affects the quality of life, and often requires reduction or suspension of chemotherapy and/or radiotherapy, thereby decreasing the relative dose intensity, which may worsen prognosis (Shumsky et al., 2019).

Benzydamine hydrochloride is a widely used drug in dentistry , a non-steroidal anti-inflammatory drug, has shown topical anti-inflammatory, analgesic, anaesthetic and antimicrobial effects and is used to attenuate inflammatory conditions like radiation -induced oral mucositis or chemotherapy-induced oral mucositis (Nithin, et al.,2018). In addition to this, Benzydamine HCL is available on the Egyptian market and its price is economical .Rebamipide is a drug used for the treatment of gastritis and gastric ulcer. The mechanisms involved in the anti-ulcer and cytoprotective effects of rebamipide have been reported to include an effect on prostaglandin E2 synthesis via COX-2 expression (Udagawaet al ., 2003), up-regulation of growth factors and their receptors such as EGF and HGF ,induction of mucus secretion ,anti-free radical effects and inhibition of the production of inflammatory cytokines such as IL-1, IL-8, and TNF-α (Yasuda et al., 2011).

Different treatment options and drugs have been tested in OM, only some of which exhibited clinical relevance such as oral cryotherapy, keratinocyte growth factor and amino acids enriched diets. Therefore, there is a clear requirement for new approaches to the prevention and effective treatment of OM (Mallick, Benson, & Rath, 2016)

In 2019 a meta-analysis performed by Akagi and his colleagues (Akagi et al., 2019) showed that gargling treatment with Rebamipide is superior to placebo for the development of mucositis and stomatitis due to chemo-radio-therapy, especially for severe cases of Grade 3 or higher. However, in order to confirm these trials, further well-designed analyses are needed, and evaluation of adverse events in observational studies are also required.

ELIGIBILITY:
Inclusion Criteria:Male and female patients with head and neck cancer and who will be prescribed radiotherapy at least 60 Gy (Roopashri et al., 2011).

* Patients who will sign an informed consent,
* Patients older than 18 years of age,
* Patients having normal renal and liver functions

Exclusion Criteria:• . Use of dentures, or having any source of infection in the mouth.

* Allergy to rebamipide or benzydamine hydrochloride(Nithin et al., 2018) .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of oral mucositis | 6-8 week will evaluate patient weekly from start of radiation
  The following parameters will be recorded at baseline , every week from start of radiation therapy and 2 weeks after end of RT . The patient will be visited once prior to radiation then weekly throughout the period of the study:1-WHO Mucositis scale (Organization, 1979),Oral Mucositis Assessment Scale (OMAS)(Sonis, 2004)

SECONDARY OUTCOMES:
The pain score | 8 week
  The pain score (Cella et al., 2003) :will recorded using a 10-point scale, the Numerical Rating Scale (NRS), wherein 0=no pain and 10=worst possible pain
  . These objective assessments will be obtained weekly following initiation of radiotherapy (4-6 week ) and until 2 weeks after end of RT .

CONTACTS AND LOCATIONS:
Overall Officials: souheir Jafar, professor, Study Director — Cairo University
Locations (1):
- Kasr El-Einy Center of Radiation Oncology and Nuclear Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data collection and storage will be the responsibility of the candidate. Patient's personal information will be available to the candidate only. While the clinical and analytical data will be available to the entire research team.

REFERENCES:
- [Derived] Elsaadany B, Anayb SM, Mashhour K, Yossif M, Zahran F. Rebamipide gargle and benzydamine gargle in prevention and management of chemo-radiotherapy and radiotherapy-induced oral mucositis in head and neck cancer patients (randomized clinical trial). BMC Oral Health. 2024 Jun 1;24(1):645. doi: 10.1186/s12903-024-04379-3. PMID 38824583